CLINICAL TRIAL: NCT02288026
Title: Comparison of Different Types of Surgery in Treating Patients With Early-stage Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other); Beijing Chest Hospital (Other); Beijing Tongren Hospital (Other); Peking University First Hospital (Other); China-Japan Friendship Hospital (Other); Peking Union Medical College Hospital (Other); Chinese PLA General Hospital (Other); Beijing Anzhen Hospital (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xiuyi zhi, Chief Physician, Xuanwu Hospital, Beijing
Other Study IDs: D14110700020000
Record Dates: First submitted 2014-10-11; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Stage IA Non-small Cell Lung Cancer; Adenocarcinoma of the Lung; Squamous Cell Lung Cancer
Keywords: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma, Bronchogenic; Bronchial Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Lung Neoplasms; Carcinoma, Bronchogenic; Bronchial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Arm I: Patients undergo lobectomy
- Arm II: Patients undergo a wedge resection or anatomical segmentectomy

SUMMARY:
The purpose of this study is to compare early-stage peripheral non-small cell lung cancer lobectomy and sub-lobectomy surgery to evaluate if sub-lobectomy is as feasible and effective for the treatment of early-stage (diameter ≤2cm) peripheral non-small cell lung cancer as lobectomy.

DETAILED DESCRIPTION:
Objectives:To establish a database of patients with early lung cancer surgery,and evaluate if sub-lobectomy surgery is as feasible and effective as lobectomy surgery in patients with early-stage peripheral non-small cell lung cancer,by assessing the retainability of lung function.and improvement of quality of life in those patients.

Outline:This is a prospective, matched, controlled, open, multi-center clinical study. Select the early-stage peripheral NSCLC 630 patients (diameter≤2cm), according to age and lesion type (GGO component ratio) two matching factor of 1: 2 assigned to sub-lobectomy group and lobectomy group.Patients are followed up every 3 months for the first year and then every 6 months for the other 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. clinically diagnosed with stage I peripheral non-small cell lung cancer suitable for lobectomy.
2. T≤2cm，N0，M0.
3. aged 60 to 80 years old.
4. ECOG≤2.
5. according to the Ministry of Health, "with primary lung cancer diagnostic and treatment practices" (2011 edition) completed preoperative clinical staging examination.
6. voluntary participation, signed informed consent.

Exclusion Criteria:

1. pathologic stage is N1, N2, or M1a.
2. received postoperative adjuvant therapy (chemotherapy or targeted therapy).
3. radiotherapy or chemotherapy before surgery.
4. small cell lung cancer
5. benign lesions
6. patient unwilling to cooperate with surgery or observation.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are stratified according to age and lesion type (GGO component ratio) two matching factor of 1: 2 to the lobectomy and sub-lobectomy surgery groups.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | participants will be followed from surgical treatment at least 5 years unless any evidence of disease progression or death

SECONDARY OUTCOMES:
Overall survival | at least 5 years
Pulmonary function | Forced expiratory volume in one second, FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Xiuyi Zhi, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu hospital capital medical university, Beijing, China